CLINICAL TRIAL: NCT04271930
Title: Mindfulness Meditation and Sleep Disturbances in Hematopoietic Cell Transplant Patients: Inflammatory Mechanisms
Brief Title: Effect of Sleep Quality on Hematopoietic Cell Transplant Patient Outcomes
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: This study terminated early due to lack of participant retention
Sponsor: Medical College of Wisconsin (Other)
Responsible Party: Principal Investigator, Jennifer M. Knight, Assistant Professor, Medical College of Wisconsin
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: PRO00036928
Record Dates: First submitted 2020-02-14; First posted 2020-02-17 (Actual); Last update posted 2024-10-09 (Actual); Status verified 2024-10

CONDITIONS: Sleep; Multiple Myeloma
Keywords: Sleep; Insomnia; Mindfulness Awareness Practices for Insomnia; Sleep Health Education; Multiple Myeloma; Autologous Hematopoietic Cell Transplantation; Depression; Inflammation; Sleep hygiene; Fatigue
MeSH Terms: conditions — Multiple Myeloma; Sleep Initiation and Maintenance Disorders; Depression; Inflammation; Sleep Hygiene; Fatigue

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Mindfulness Awareness Practices for Insomnia (Experimental): Participants will be instructed to practice mindfulness techniques on a daily basis, beginning with 5 minutes and increasing to 20 minutes over the course of the 6-week intervention - as is standard with the Mindfulness Awareness Practices (MAPs) course - with practice prior to bedtime. An intervention training manual is the cornerstone of standardized delivery of MAP-I. Participants are also provided with a book on mindfulness (Fully Present: The Science, Art, and Practice of Mindfulness, authored by the Mindfulness Awareness Research Center (MARC) leader and MAP-I instructor Diana Winston) as well as access to the University of California Los Angeles (UCLA) Mindful App courtesy of the MARC at UCLA (via personal iPhone or study-administered tablets per patient preference), which contains pre-recorded guided meditations for use in daily practice.
  Interventions: Behavioral: Mindfulness Awareness Practices for Insomnia
- Sleep Health Education (Active Comparator): Six individual 1-hour videos will be shown to participants at the same time points as, and with equal duration to, the MAP-I intervention. These videos will be recorded presentations that have been modified for HCT recipients based upon similar SHE interventions delivered in prior studies. Similar to the intervention group, patients in the SHE group will also participate in group Zoom chat sessions with equal frequency and duration lead by a study research coordinator. These sessions will allow for general patient interaction to discuss sleep and any questions or comments they may have, as lead by the group facilitator.
  Interventions: Behavioral: Sleep Health Information

INTERVENTIONS:
Behavioral: Mindfulness Awareness Practices for Insomnia — MAP-I is a curriculum-based intervention that incorporates practice prior to bed, use of practice in the bed during night-time awakenings, and daily body scan.
  Arms: Mindfulness Awareness Practices for Insomnia
Behavioral: Sleep Health Information — A video SHE seminar will serve as active comparator for nonspecific treatment elements that pose rival explanations for the effectiveness of MAP-I.
  Arms: Sleep Health Education

SUMMARY:
This randomized, controlled study will compare Mindfulness Awareness Practices for Insomnia (MAP-I) to sleep health education (SHE) in subjects receiving autologous hematopoietic cell transplant for multiple myeloma.

DETAILED DESCRIPTION:
This randomized controlled study will evaluate the feasibility of implementing a mindfulness intervention targeting inpatient autologous hematopoietic cell transplantation (HCT) recipients (first HCT) with multiple myeloma (MM) and the preliminary efficacy of Mindfulness Awareness Practices for Insomnia (MAP-I) vs. sleep health education (SHE) to improve insomnia outcomes, cellular and transcriptomic markers of inflammation, and insomnia associated behavioral symptoms (depression, fatigue).

Patients enrolled in this study will be randomized to either receive MAP-I or SHE starting 2-4 weeks prior to HCT. Patients will receive two sessions prior to inpatient admission for HCT, and four sessions in the two weeks of hospitalization following HCT, for a total of six intervention (or control) sessions.

Primary Objective: Determine the feasibility of implementing MAP-I among HCT recipients under first autologous HCT for MM.

ELIGIBILITY:
Inclusion Criteria:

* ≥18 years of age
* ≤ 1 year since initiation of systemic anti-myeloma therapy
* No prior progression or relapse of myeloma prior to HCT
* Patient should be eligible to receive melphalan 200 mg/m2 as conditioning regimen
* Stem cell graft with > 2.0 x10^6 cluster of differentiation 34 cells (CD34+)/kg available for transplant
* Karnofsky Performance Score (KPS) ≥70
* Agreeable to random assignment and data collection, including survey completion and blood draws
* Available to attend the outpatient intervention portion.
* Voluntary written consent must be given before performance of any study related procedure not part of standard medical care, with the understanding that consent may be withdrawn by the subject at any time without prejudice to future medical care

Exclusion Criteria:

* Prior autologous HCT
* Outpatient HCT
* Presence of coexistent amyloidosis
* Presence of known Obstructive Sleep Apnea (OSA)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 24 (Actual)
Dates: Start 2020-11-01 (Actual); Primary Completion 2023-05-23 (Actual); Study Completion 2023-05-23 (Actual)

PRIMARY OUTCOMES:
Number of Participants Enrolling in the Study | Up to 2 weeks
  This outcome measure is the number of participants signed consent and were enrolled compared to the number of potential participants assessed for eligibility.
Number of Participants Completing Study Procedures | 100 days after transplant procedure
  This outcome measure is the number of participants completing the required study procedures compared to the number of participants initiating study procedures.

CONTACTS AND LOCATIONS:
Overall Officials: Jennifer Knight, MD, Principal Investigator — Medical College of Wisconsin
Locations (1):
- Froedtert Hospital and the Medical College of Wisconsin, Milwaukee, Wisconsin, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Henley EC, Liphart HA, Morris KJ, Awoyinka I, Irwin MR, Costanzo ES, Winston D, D'Souza A, Stolley M, Dhakal B, Mohan M, Pasquini MC, Cole SW, Doerwald ES, Bendis PC, Rentscher KE, Rumble ME, Szabo A, Rao S, Knight JM. Mindfulness vs. sleep education during autologous hematopoietic cell transplantation for multiple myeloma: Feasibility of a randomized controlled pilot study. Contemp Clin Trials Commun. 2025 Aug 18;47:101540. doi: 10.1016/j.conctc.2025.101540. eCollection 2025 Oct. PMID 40893725